CLINICAL TRIAL: NCT05661136
Title: Maternal Postoperative Temperature After Cesarean Delivery Under Spinal Anesthesia With Warmed Intravenous Fluids: Randomized Controlled Trial With Versus Without Lower Body Forced Air Warming
Brief Title: Maternal Postop Temperature After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CTIL - 0562-22-TLV -
Record Dates: First submitted 2022-12-06; First posted 2022-12-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Temperature Change, Body; Cesarean Delivery; Spinal Anesthesia
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: two arms: lower body forced air warming versus none
Who Masked: Outcomes Assessor
Masking Description: Postanesthesia care unit nurses assess primary outcome and will not know the group assignment
  Sample size was calculated for the primary outcome of difference between the groups in maternal temperature on arrival to the post-anesthesia care unit. We calculated the a priori sample size, WinPepi, based upon a prior publication that compared Active-Warming versus No-Warming, mean(standard deviation) 35.9(0.5)0 C versus 35.5(0.5), power 90%, 0.05 two-sided significance (Cobb et al). For clinical significance we calculated sample size with a mean difference of 0.50 C, with SD 0.5, power 90%, two sided significance with potential for 10% dropouts, total 66 women, 33 per group, and without dropouts, 22 per group total 44 women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm air blower (Experimental): Intra-operative lower-body forced-air warming after spinal anesthesia and co-loading 1000 mL liters of IV warmed-fluids started prior to performing spinal anesthesia
  Interventions: Device: Warm air blower
- Control (Active Comparator): Co-loading of 1000 mL liters of IV warmed-fluids started prior to performing spinal anesthesia
  Interventions: Other: Control: Lower body blanket not attached to warm air blower

INTERVENTIONS:
Device: Warm air blower — Lower body blanket with warm air blower set at 44 deg c started after spinal anesthesia when patient placed in supine/left lat position
  Arms: Warm air blower
Other: Control: Lower body blanket not attached to warm air blower — Control: Lower body blanket placed, not attached to warm air blower
  Arms: Control

SUMMARY:
It is unclear whether routine addition of intra-operative forced-air warming in addition to warmed intravenous fluids during cesarean delivery under spinal anesthesia is beneficial. In this single-center randomized trial, we aim to test the primary null hypothesis that our current protocol of warmed intravenous fluids is similar to a combination of warmed intravenous fluids with intra-operative lower-body forced-air warming to maintain maternal temperature after cesarean delivery under spinal anesthesia.

We also aim to assess the rate of maternal shivering during and after the procedure between the two groups, the maternal thermal comfort score, neonatal Apgar scores and umbilical pH levels. If we demonstrate no clinically important difference between the two interventions, clinicians will be able to continue our current protocol of warmed intravenous fluids only during cesarean delivery.

DETAILED DESCRIPTION:
Primary aim Investigate whether a combination of intra-operative lower-body forced-air warming and warmed IV fluids is superior to our current standard of warmed IV fluids alone in influencing maternal core temperature following spinal anesthesia for cesarean delivery.

Secondary aim

1. To compare mean core temperature on arrival to post-anesthesia care unit (PACU) in women who received combination of intra-operative lower-body forced-air warming and warmed IV fluids versus IV fluids alone
2. To compare incidence of hypothermia among women who received combination of intra-operative lower-body forced-air warming and warmed IV fluids versus IV fluids alone
3. To compare incidence of shivering following recovery in post anesthesia care unit (PACU) in women who received combination of intra-operative lower-body forced-air warming and warmed IV fluids versus IV fluids alone
4. To compare thermal comfort levels for women who received combination of intra-operative lower-body forced-air warming and warmed IV fluids versus IV fluids alone
5. To compare use of meperidine in post anesthesia care unit (PACU) to treat postoperative shivering, in women who received combination of intra-operative lower-body forced-air warming and warmed IV fluids versus IV fluids alone
6. To compare newborn outcomes (rectal temperature at birth, umbilical vein pH & Apgar scores post-delivery) in women who received combination of intra-operative lower-body forced-air warming and warmed IV fluids versus IV fluids alone

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age between 18-50 years old
3. American Society of Anesthesiologists (ASA) physical status 2-3
4. Gestational age greater than 37 completed weeks
5. Singleton pregnancy
6. Elective cesarean delivery.

Exclusion Criteria:

1. Known allergy to local anesthetics
2. Contraindication for spinal anesthesia

   1. Patient refusal
   2. Bleeding diathesis
   3. Neuropathy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
The mean core temperature | baseline, immediately before spinal anesthesia, 60 minutes following spinal anesthesia and then every 30 minutes for 2 hours (last measurement prior to discharge)
  The primary aim is the mean core temperature on arrival to PACU. The means for the two groups will be compared.

SECONDARY OUTCOMES:
Maternal hypothermia | 60 minutes following spinal anesthesia
  Maternal hypothermia yes/no defined as core body temperature <36°C
Shivering | Postoperative - every 30 minutes for 2 hours (last measurement prior to discharge)
  Shivering score - 0 - no shivering
  1. - One or more of the following: piloerection, peripheral vasoconstriction, peripheral cyanosis without other cause, but without visible muscular activity
  2. - Visible muscular activity confined to one muscle group
  3. - Visible muscular activity in more than one muscle group
  4. - Gross muscular activity involving the whole body
Maternal thermal comfort | baseline, immediately before spinal anesthesia , 60 minutes following spinal anesthesia, and then every 30 minutes for 2 hours (last measurement prior to discharge)
  Maternal thermal comfort scores (• Thermal comfort scale - a 0 to 10 scale will be used with the descriptors to a single question - "How warm or cold are you?
  o "Worst imaginable cold", " thermally neutral, " and " insufferably hot " representing the 0, 5, and 10 of the scale, respectively) will be obtained at baseline, 30 minutes during surgery, and on admission to PACU
Meperidine | Postoperative - up to two hours during PACU recovery after the procedure
  Meperidine administration (timing and dose) used to treat shivering
Apgar | 1 and 5 minutes after newborn delivery
  Apgar scores (at 1 and 5 minutes) will be determined by the pediatrician (not involved in the study)
Newborn Temperature | Upon newborn's arrival to newborn ward - approximately 30 minutes following delivery
  Newborn rectal temperature
Umbilical vein pH | Immediately following placenta removal intraoperatively
  venous blood gases will be obtained for analysis from a double-clamped segment of umbilical cord

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv SMO, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
no plan